CLINICAL TRIAL: NCT04421950
Title: Plasma and Urine Profiles of Blueberry Derived Polyphenols After a Short Term Intervention With Blueberry in Children With Typical Low Fruit and Vegetable Consumption.
Brief Title: The Blueberry Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 260493; 6026-51000-012-06S (Other Grant/Funding Number: USDA-ARS); P20GM109096 (NIH)
Record Dates: First submitted 2020-05-26; First posted 2020-06-09 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded randomized control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wild Blueberry Supplement (Active Comparator): 30 grams of wild blueberry powder per day in foods items provided to them
  Interventions: Dietary Supplement: Wild blueberry containing foods
- Placebo supplement (Placebo Comparator): Food items will be provided to them without the wild blueberry power.
  Interventions: Dietary Supplement: Placebo containing foods

INTERVENTIONS:
Dietary Supplement: Wild blueberry containing foods — Foods that contain wild blueberry supplement to deliver up to 30 grams of blueberry powder
  Arms: Wild Blueberry Supplement
Dietary Supplement: Placebo containing foods — Foods that do not contain the blueberry powder but a placebo
  Arms: Placebo supplement

SUMMARY:
This is a research study about the effects of blueberries on the health of children who do not eat much fruits and vegetables. By doing this study, we hope to find out what nutrients from blueberries appear in the blood and urine of the child

DETAILED DESCRIPTION:
This is a double blinded randomized control trial aiming to characterize the profile of polyphenol-derived metabolites in plasma and urine for children ages 11-12 years supplemented short term with wild blueberry powder. The study will assess if a short-term supplementation (5 days) with wild blueberry powder impacts immune responses as well as markers for cardiovascular and bone health. Up to 44 children will be recruited. The participants will attend three visits at Arkansas Children's Nutrition Center.

ELIGIBILITY:
Inclusion Criteria:

* Eats <1.5 cup of fruit and <2.0 cup of vegetables per day
* Boys or girls
* All ethnicities
* All BMIs

Exclusion Criteria:

* Known allergy to blueberries
* Epilepsy
* Asthma
* Chronic kidney disease
* Hormonal disease
* Autoimmune disease
* Bleeding disorders
* Chronic infections
* Type 2 and Type 1 diabetes mellitus
* Attention deficit hyperactivity disorder
* Opposition defiant disorder
* Autistic spectrum disorder
* Pre-existing medical conditions or medications as determined by the investigators to affect the outcomes of interest
* If the participants/parents perceive barriers with adhering to low-polyphenol meals
* Parent or child refusal to stop nutritional supplements
* Parent or child refusal to have blood drawn

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Diaz, MD, Principal Investigator — Arkansas Children's Reserach Institute
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-four children were enrolled at the Arkansas Children's Nutrition Center, with the first participant enrolled on April 23, 2021, and the last participant on August 4, 2022
Pre-assignment Details: After enrollment, the children were placed on a low-polyphenol diet for 48 hours. Following this period, they were assigned to consume either wild-blueberry products (n = 22) or placebo-containing products (n = 22).
Groups:
- Wild Blueberry Supplement: 30 grams of wild blueberry powder per day in food items provided to participants
  Wild blueberry containing foods: Foods that contain wild blueberry supplement to deliver up to 30 grams of blueberry powder
- Placebo Supplement: Food items were provided to study participants without the wild blueberry power.
  Placebo containing foods: Foods that do not contain the blueberry powder but a placebo
Period: Overall Study
Arm/Group | Wild Blueberry Supplement | Placebo Supplement
Started | 22 | 22
Completed | 18 | 20
Not Completed | 4 | 2
Not completed — Dropped or lost to follow up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Wild Blueberry Supplement: 30 grams of wild blueberry powder per day in foods items provided to study participants
  Wild blueberry containing foods: Foods that contain wild blueberry supplement to deliver up to 30 grams of blueberry powder
- Placebo Supplement: Food items without wild blueberry power were provided to study participants.
  Placebo containing foods: Foods that do not contain the blueberry powder but a placebo
- Total: Total of all reporting groups
Arm/Group | Wild Blueberry Supplement | Placebo Supplement | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.94 (0.60) | 11.94 (0.60) | 11.94 (0.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was assessed per NIH criteria
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 4 | 6
    White | 18 | 16 | 34
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 44
BMI percentile [Mean (Standard Deviation); unit: percentile] — Anthropometric measurements, including body weight and height, were obtained using standardized techniques, with the children wearing light clothing and no shoes. All measurements were taken in duplicate, or in triplicate if the initial measures did not meet acceptable agreement. Age-, sex-, and height-specific body mass index percentiles were calculated using growth charts from the CDC.
  percentile | 72.2 (30.6) | 50.7 (30.6) | 63.5 (32.9)
Systolic blood pressure percentile [Mean (Standard Deviation); unit: percentile] — Blood pressure was measure following the 2017 guidelines from the American Academy of Pediatrics. Blood pressure percentiles were calculated using reference standards to allow comparisons across children of all ages, heights, and sex.
  percentile | 45 (27) | 48 (29) | 47 (28)
Diastolic blood pressure percentile [Mean (Standard Deviation); unit: percentile] — Blood pressure was measure following the 2017 guidelines from the American Academy of Pediatrics. Blood pressure percentiles were calculated using reference standards to allow comparisons across children of all ages, heights, and sex.
  percentile | 53 (22) | 51 (20) | 52 (21)
Peak VO2 [Mean (Standard Deviation); unit: ml/kg/min] — A graded exercise test was performed to determine peak oxygen uptake (peak VO2). A bicycle fitness test was conducted, during which the resistance of the stationary bicycle was gradually increased. The children were told that they could stop the test at any time if they did not wish to continue but were encouraged to perform maximally. During the test, the children wore an indirect calorimetry face mask to assess their oxygen uptake (VO2), carbon dioxide production (VCO2), and respiratory exchange ratio (RER; VCO2/VO2).
  Peak VO2 (ml/min) was normalized per body weight.
  ml/kg/min | 33.1 (9.4) | 35.9 (10.9) | 34.5 (10.2)
Flow mediated dilation of the brachial artery [Mean (Standard Deviation); unit: Percentage of artery diameter] — Endothelial function was measured during visits #2 using ultrasound (GE Vivid 7 Ultrasound system with 5.0-13.0 MHz linear transducer, GE Healthcare, Chicago, IL, USA) to assess brachial artery flow-mediated dilation (FMD). This technology used sound waves (ultrasound) to visualize the diameter of the brachial artery. A baseline image of the brachial artery was recorded at rest. Population: Flow mediated dilation of the brachial artery (%, FMD) were taken at visit 2 before the participants received the study products. Six participants dropped out of the study or were lost to follow-up by visit 2. Additionally, two FMD measurements were either unsuccessful or did not meet the quality criteria for inclusion in the analysis, resulting in a total of 36 baseline FMDs. There are currently no reference standards for FMD in children.
  Percentage of artery diameter
    number analyzed (Participants) | 16 | 20 | 36
    (all) | 11.8 (4.2) | 11.6 (4.8) | 11.6 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Phenolic Acid Metabolites Measured in Plasma and Urine After Dietary Intervention
Description: Fasting Blood and urine were collected at visit two and three following an overnight fasting. At visit three, children consumed a single dose of the study product and plasma and urine were collected
Time Frame: Measurements were conducted hourly for 5 hours; the cumulative number of metabolites characterized over the 5 hours is reported
Population: Phenolic-derived metabolites were characterized in the samples using an ultra-high performance liquid chromatography method coupled with mass-spectrometry/mass spectrometry multiple reactions monitoring
Measure: Number; unit: Counts of metabolites
Groups:
- Wild Blueberry Supplement: 30 grams of wild blueberry powder per day in foods items were provided to study participant
  Wild blueberry containing foods: Foods that contain wild blueberry supplement to deliver up to 30 grams of blueberry powder
- Placebo Supplement: Food items without the wild blueberry power were provided to study participants,
  Placebo containing foods: Foods that do not contain the blueberry powder but a placebo
Arm/Group | Wild Blueberry Supplement | Placebo Supplement
Number analyzed (Participants) | 18 | 20
Counts of metabolites
  Plasma | 13 | 0
  Urine | 25 | 3

2. Secondary Outcome: Number and Percentage of Lymphocytes Cluster of Differentiation 4 (CD4), Lymphocytes Cluster of Differentiation 8 (CD8) and Natural Killer (NK) Cells
Description: Mitogen stimulated blood will be stained with combinations of fluorochrome-labeled antibodies and analyzed by flow cytometry. Absolute and relative number of CD4, lymphocytes CD8 and natural killer (NK) will be compared between groups.
Time Frame: up to 2 weeks
Reporting Status: Not Posted

3. Secondary Outcome: T-lymphocyte Responsiveness to Immune Stressors
Description: Blood will be collected following an overnight fast after 5 days on the intervention. Whole blood will be cultured and cells stressed with E. coli lipopolysaccharide (LPS) to induce cytokine release from immune cells. Cytokines will be assayed using electrochemiluminescence based detection platform with multiplexed immunoassays, and their levels compared between study groups.
Time Frame: up to 2 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Endothelial Function by Brachial Artery Flow Mediated Dilation
Description: Endothelial-dependent flow-mediated vasodilation of the brachial artery in the fasting state was measured using high resolution ultrasound at enrollment and after 5 days on the intervention. This technology uses sound waves (ultrasound) to visualize the diameter of the brachial artery. A baseline image of the brachial artery will be recorded at rest. A blood pressure cuff will be placed around the lower arm and the cuff will be inflated to 50 mmHg above systolic pressure for 5 minutes, followed by rapid deflation of the cuff. The diameter of the brachial artery will be measured from ultrasound images captured throughout the 8 minute recording protocol. The percent change in the brachial artery will be compared between and within groups.
Time Frame: up to 2 weeks
Measure: Mean (Standard Deviation); unit: percentage change in arterial diameter
Groups:
- Placebo Supplement: Food items without the wild blueberry power were provided to study participants
  Placebo containing foods: Foods that do not contain the blueberry powder but a placebo
Arm/Group | Wild Blueberry Supplement | Placebo Supplement
Number analyzed (Participants) | 18 | 20
percentage change in arterial diameter | 9.4 (3.4) | 9.4 (3.0)
Statistical Analysis 1: Comparison: Wild Blueberry Supplement vs Placebo Supplement; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Arm/Group | Wild Blueberry Supplement | Placebo Supplement
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 2/22 | 2/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wild Blueberry Supplement (N=22) | Placebo Supplement (N=22)
High blood pressure (General disorders) | 2 (2) | 2 (2) — Blood pressure marked as elevated
Gastrointestinal symptoms (Gastrointestinal disorders) | 1 (1) | 1 (1) — Nausea and / or vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT04421950/Prot_SAP_000.pdf